CLINICAL TRIAL: NCT00088985
Title: Phase II Trial Evaluating The Efficacy Of A Multiepitope Dendritic Cell Vaccine Given With Trastuzumab And Vinorelbine For The Treatment Of Women With Metastatic Breast Cancer That Express HLA-A0201
Brief Title: Vaccine Therapy, Trastuzumab, and Vinorelbine in Treating Women With Locally Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0310; P50CA058223 (NIH); R21CA105837 (NIH); KG100307 (Other Grant/Funding Number: Susan G Komen for the Cure)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Cell Vaccine (Experimental): Dendritic Cells: Dosage: 20 x 106 dendritic cells (DCs) given per treatment Vinorelbine:25 mg/m2 will be administered i.v biweekly Trastuzumab: 6mg/Kg administered by i.v. biweekly
  Interventions: Biological: therapeutic autologous dendritic cells; Biological: trastuzumab; Drug: vinorelbine ditartrate

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells — 10 μg/kg subcutaneously (sc) each day for four days or g-CSF at 5 μg/kg sc each day for four days with GM-CSF 250 μg/m2 sc each day for four days. G-CSF and/or GM- CSF will be self-administered. On the fifth day patients will have two intravenous lines placed in the apheresis area of the Blood Bank and then undergo a 15 litre apheresis collection
Biological: trastuzumab — 4 mg/kg intravenously, every 14 days
Drug: vinorelbine ditartrate — Vinorelbine 25 mg/m2 will be administered intravenously, every 14 days

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with monoclonal antibody therapy and chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with trastuzumab and vinorelbine works in treating women with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of multiepitope autologous dendritic cell vaccine, trastuzumab (Herceptin^®), and vinorelbine by measuring the change in the largest dimension of metastatic lesions, in women with locally recurrent or metastatic breast cancer that does not overexpress human epidermal growth factor receptor 2 (HER2)/neu.

Secondary

* Determine the ability of this regimen to induce functional antigen-specific T cells in these patients by measuring ex-vivo antigen-specific T-cell activity against peptide-pulsed dendritic cells and tumor targets by tetramer staining and intracellular cytokine assays.

OUTLINE:

* Autologous dendritic cell mobilization and harvest: All patients undergo autologous dendritic cell mobilization with filgrastim (G-CSF) and/or sargramostim (GM-CSF) subcutaneously daily for 4 days followed by apheresis. Mobilized peripheral blood is processed for the production of dendritic cells by cluster of differentiation (CD)34-positive cell selection. The dendritic cells are expanded and then pulsed with E75 and E90 peptides.
* Treatment: Patients receive vinorelbine IV over 6-10 minutes and trastuzumab (Herceptin ^®) IV over 90 minutes on day 1. Patients also receive autologous dendritic cells pulsed with E75 and E90 peptides subcutaneously over 2-5 minutes on day 1*. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Note: *If treatment is given locally, the vaccine therapy will be given at University of North Carolina (UNC) -Chapel Hill the following day.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Locally recurrent or metastatic disease
* HLA-A0201 positive by DNA genotyping
* HER2/neu expression at least 1+ by immunohistochemistry of tumor sample
* Central Nervous System (CNS) metastases allowed provided on therapy for 3 months and stable
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hematocrit > 33%

Hepatic

* Transaminases ≤ 3 times upper limit of normal
* Bilirubin ≤ 2 times normal
* Hepatitis B surface antigen negative

Renal

* Creatinine < 2.0 mg/dL

Cardiovascular

* Ejection fraction > 45% by multigated acquisition scan (MUGA) OR
* Left ventricular function normal by echocardiogram
* No serious cardiac condition that would preclude study participation or compliance

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No serious medical or psychiatric condition that would preclude study participation or compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed

Chemotherapy

* More than 30 days since prior cytotoxic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* More than 30 days since prior hormonal therapy
* No concurrent hormonal therapy
* No concurrent systemic steroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent bisphosphonates for bone metastases allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Serody, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 patients enrolled; 23 were human leukocyte antigen (HLA:A2) negative, 11 withdrew/refused treatment prior to start, 4 consented/not treated due to study closure, 3 went to a different study, 2 died before treatment, 2 were human epidermal growth factor receptor 2 (HER-2/neu) not detectable, and 4 patients ineligible. 7 patients were evaluable.
Groups:
- Dendritic Cell Vaccine: Dendritic Cells (DCs): Dosage: 20 x 106 DCs given per treatment Vinorelbine:25 mg/m2 will be administered i.v biweekly Trastuzumab: 6mg/Kg administered by i.v. biweekly
  therapeutic autologous dendritic cells: 10 μg/kg subcutaneously (sc) each day for four days or g-CSF at 5 μg/kg sc each day for four days with Granulocyte-macrophage colony-stimulating factor (GM-CSF) 250 μg/m2 sc each day for four days. G-CSF and/or GM-CSF will be self-administered. On the fifth day patients will have two intravenous lines placed in the apheresis area of the Blood Bank and then undergo a 15 litre apheresis collection
  trastuzumab: 4 mg/kg intravenously, every 14 days
  vinorelbine ditartrate: Vinorelbine 25 mg/m2 will be administered intravenously, every 14 days
Period: Overall Study
Arm/Group | Dendritic Cell Vaccine
Started | 7
Completed | 4
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Dendritic Cell Vaccine: Dendritic Cells: Dosage: 20 x 106 DCs given per treatment Vinorelbine:25 mg/m2 will be administered i.v biweekly Trastuzumab: 6mg/Kg administered by i.v. biweekly
  therapeutic autologous dendritic cells: 10 μg/kg subcutaneously (sc) each day for four days or g-CSF at 5 μg/kg sc each day for four days with GM-CSF 250 μg/m2 sc each day for four days. G-CSF and/or GM- CSF will be self-administered. On the fifth day patients will have two intravenous lines placed in the apheresis area of the Blood Bank and then undergo a 15 litre apheresis collection
  trastuzumab: 4 mg/kg intravenously, every 14 days
  vinorelbine ditartrate: Vinorelbine 25 mg/m2 will be administered intravenously, every 14 days
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 64.43 [54 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response measured by Response Evaluation Criteria In Solid Tumors (RECIST), (Complete Response + Partial Response)
  Complete Response (CR)- Disappearance of all target lesions
  Partial Response (PR)-at least a 30% decrease in the longest diameters of target lesions, taking as reference the baseline longest diameter.
Time Frame: 6 months following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Immune Response
Description: Measured by intracellular cytokine staining for Interferon-gamma (INFgamma) and cluster of differentiation (CD107) up regulation and tetramer. A fourfold increase in the number of cluster of differentiation (CD8+) tetramers comparing prevaccine with peak postvaccine values indicated an immune response to the therapy.
Time Frame: 3 months following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 7
Participants
  CD8+ Tetramer Increased | 7
  No Change | 0

ADVERSE EVENTS:
Time Frame: Toxicity was assessed on day 14 of each cycle and again 15-30 days post treatment.
Arm/Group | Dendritic Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dendritic Cell Vaccine (N=7)
Fever (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dendritic Cell Vaccine (N=7)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Edema (General disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 3
Headache (Nervous system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Leukocytes (total WBC) (Investigations) | 3
Lymphopenia (Investigations) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain - Other (Specify) (General disorders) | 1 — wrist pain
Platelets (Investigations) | 1

LIMITATIONS AND CAVEATS:
Study was terminated due to unavailable funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes